CLINICAL TRIAL: NCT03122093
Title: Celiac Disease and Diabetes Longitudinal Follow-up and Evaluation Study (CD-LiFE)
Brief Title: Celiac Disease and Diabetes Longitudinal Follow-up and Evaluation Study
Acronym: CD-LiFE
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Farid Mahmud, Principal Investigator, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000053646
Record Dates: First submitted 2017-04-03; First posted 2017-04-20 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Celiac Disease; Celiac; Diabetes Mellitus, Type 1
Keywords: pediatric; dietary treatment; celiac disease; T1D
MeSH Terms: conditions — Celiac Disease; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CD-DIET Gluten-Free Diet Group: This former randomized control trial (RCT) group received a gluten-free education and continued support from a dietitian for a 1-year period via the CD-DIET Study (NCT01566110)
- CD-DIET Gluten-Containing Diet Group: This former RCT group did not receive a gluten-free education and 1-year support from a dietitian via the CD-DIET Study (NCT01566110), but rather a single gluten-free education session upon exiting the study.
- CD-DIET Ineligibles/Refusals: This group contains T1D/CD individuals who were not eligible or refused to join the CD-DIET RCT (e.g. already self-selected their diet or had no interest in being randomized). These individuals were instead redirected to the clinical route.

SUMMARY:
To the investigators' knowledge, no single long-term prospective observational study has assessed dietary factors, diabetes clinical variables (metabolic control and associated complications), and self -perceived health and wellness in T1D patients (both pediatric and adult) with CD identified by screening (positive/weakly positive serology). The aim of the current study is to observe the short- and long-term outcomes for Type 1 diabetic patients with new serology positive asymptomatic CD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 8 and 50 years with positive/weakly positive serologic CD screening or who have completed the CD-DIET trial.
2. Diagnosis of T1D by American Diabetes Association (ADA) criteria with duration of T1D equal to or greater than 1 year from time of signing Screening Informed Consent for CD-DIET trial.
3. Ability of the subject or a legally authorized representative to speak and read English or French.
4. Participation in the screening portion of the CD-DIET Study.

Exclusion Criteria:

1. A condition which, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with an established diagnosis of T1D and positive/weakly positive serologic CD after entering the screening portion of the CD-DIET study will be recruited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Average Daily Gluten Intake | 2 Years
  This outcome will be measured through interview/assessment data.
Celiac Dietary Adherence | 2 Years
  This outcome will be measured through the Celiac Dietary Adherence test (CDAT) questionnaire.
TTG-IgA Serology | 2 Years
  This outcome will be measured through TTG-IgA serology testing for inflammatory markers for celiac disease.

SECONDARY OUTCOMES:
Health-related Quality of Life | 2 Years
  This outcome will be measured through the self-reported Quality of Life (PedsQL) Inventory Generic Core Scale (V.4.0) with Diabetes Module (V.3.0).
Daily Activity Levels | 2 Years
  This outcome will be measured through the self-reported Habitual Activity Estimation Scale (HAES).
Self-Perceived Wellness | 2 Years
  This outcome will be measured through a self-reported Self-Perceived Wellness Scale.
Metabolic Control | 2 years
  This outcome will be measured through self-reports and lab-provided HbA1c values.
Kidney Function | 2 years
  This outcome will be measured through lab-provided Albumin/Creatinine Ratios.
Hypoglycemic episodes. | 2 years
  The frequency and severity of hypoglycemic episodes will be recorded at each clinic visit via self-report.
Presence of Type 1 Diabetes Complications | 10 years
  This outcome will be measured by monitoring the occurence of T1D health outcomes and complications over time through long-term medical record review follow-up. Complications include, but are not limited to: nephropathy, retinopathy, and cardiovascular disease in the study population.
Presence of Celiac Disease Complications | 10 years
  This outcome will be measured by monitoring the occurence of celiac disease health outcomes and complications over time through long-term medical record review follow-up. Complications include, but are not limited to: osteoporosis and malnutrition in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Farid Mahmud, MD, Principal Investigator — The Hospital for Sick Children
Locations (6):
- Canada (6):
  - McMaster University, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences, London, Ontario
  - St. Joseph's Healthcare, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario